CLINICAL TRIAL: NCT05909111
Title: MR-Only Based Adaptive External Beam Radiation Therapy of Cervical Cancer on Ethos
Brief Title: MR-Only Based Adaptive External Beam Radiation Therapy of Cervical Cancer on Ethos Therapy: Feasibility Study
Acronym: Ethos Col
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Recherche clinique (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Sponsor-Investigator, Recherche clinique, Principal Investigator, Institut Sainte Catherine
Organization: Institut Sainte Catherine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COL-ETHOS
Record Dates: First submitted 2022-08-08; First posted 2023-06-18 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Cervical Cancer; Online Adaptative Radiation Therapy; MRI
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MRI assessment during radiation therapy course (Experimental): Patients perform on MRI every week during the 5-weeks treatment
  Interventions: Diagnostic Test: Magnetic resonance imaging

INTERVENTIONS:
Diagnostic Test: Magnetic resonance imaging — MRI weekly during the radiation treatment course (5 RMI added to the standard care)

SUMMARY:
Current management of patients treated with External Beam Radiation Therapy (EBRT) for cervical cancer with a classical Image-guided Radiation Therapy (IGRT) strategy involves a complex, not entirely satisfactory, treatment workflow. Indeed, in our institution, two workflows have been designed to take into account the inter-fraction motion of cervix and uterus : an Internal Target Volume (ITV)-based approach and a plan of the day strategy requiring both several planning-CT (Computed Tomography) acquisitions with variable bladder filling.The upcoming installation of a Varian Ethos therapy system in our institution will allow us to implement a less cumbersome online adaptive radiotherapy strategy (oART), which, by conforming to the daily anatomy, will enable a reduction in the Clinical Target Volume (CTV) to Planning Target Volume (PTV) margins leading to an expected reduction in dose delivered to organs at risk (OAR) .On the other hand, MR (Magnetic Resonance)-only treatment planning is playing an increasing role in radiotherapy, notably in the treatment of prostate cancer. MR-only workflows are known (a) to provide the most reliable delineation in soft tissues and (b) to decrease spatial uncertainties by suppressing the Magnetic Resonance Imaging (MRI)-CT co-registration. Regarding the management of cervical cancer, the importance of MRI is well established and its use becomes essential. Combining a MR-only workflow with an adaptative one on the Varian Ethos system, could lead to an improved management of patients treated for cervical cancer with an expected reduction in margins and volumes treated (thanks to MRI delineation and online adaptation) and therefore a reduction of OAR toxicity. Including regular multi-parametric MR imaging during and after the course of the treatment could also provide in the future an assessment of the treatment response. One of the important challenges in developing this specific workflow is to have a reliable synthetic CT (derived from MRI) to (a) provide electron or mass density for treatment planning calculations and (b) allow accurate online repositioning/deformation with Ethos Cone Beam Computed Tomography (CBCT). The other fundamental challenge is to provide a formal assessment of the clinical benefit of introducing MR-only simulation and planning in an oART workflow.

This project aims to demonstrate the feasibility of setting up an adaptive workflow on the ETHOS platform with the sole use of MR patient image.The project is divided into two parts. The first part consists in demonstrate the feasibility of the workflow on 15 patients with cervix cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Histologically proven cervical cancer (SCC, ADK ou adenous-SCC)
* Patient for curative RTCT treatment
* FIGO/TNM Stage IB2, IIA, IIB, IIIA, IIIB with or without lymph nodes involvement
* WHO < 2
* No pregnancy
* Informed consent dated and signed
* Patient affiliated or beneficiary of a social security scheme
* Free, informed and written consent signed by the participant and the investigator (at the latest on the day of inclusion and before any examination required by the research).

Exclusion Criteria:

* Metastatic disease
* Contraindications to IRM examinations (claustrophobia, presence of metallic elements..)
* Signes of active infection or serious health problems
* Historic of abdominal or pelvis RT
* Surgical history: partial or total hysterectomy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Tumor regression assessment CBCT | 18 months
  Volume Tumor regression on CBCT
Tumor regression assessment MRI | 18 months
  Volume Tumor regression on MRI

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Sainte Catherine, Avignon, France

IPD SHARING:
Plan to Share IPD: No